CLINICAL TRIAL: NCT05828238
Title: PET Imaging Explores the Role of SF-DEVD-2 in Monitoring Tumor Efficacy
Brief Title: Positron Emission Tomograph(PET) Imaging Explores the Role of SF-DEVD-2 in Monitoring Tumor Efficacy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, Chunjing Yu, Director, Affiliated Hospital of Jiangnan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LS2023012
Record Dates: First submitted 2023-04-11; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer Stage II; Breast Cancer Stage III; Solid Tumor
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]SF-DEVD-2 (Experimental)
  Interventions: Drug: [18F]SF-DEVD-2; Drug: [18F]-FDG

INTERVENTIONS:
Drug: [18F]SF-DEVD-2 — Patients will receive a tracer dose of 18F (2-4mCi) labelled SF-DEVD-2
Drug: [18F]-FDG — Patients will receive a tracer dose of 18F (5-10mCi) labelled FDG

SUMMARY:
This is a single arm study to determining the value of apoptotic molecular probe SF-DEVD-2 in the early evaluation of tumor efficacy and comparing it head-to-head wihe 18F-FDG(18F-2-fluoro-2-deoxy-D-glucose)

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily signed informed consent;
2. Age18-70, male or female;
3. Diagnosed with stage 2 or 3 breast cancer
4. Solid tumors、masses larger than 2cm with lymph node metastasis
5. Pathology is HER3+、triple negative patients
6. Patients to be treated with neoadjuvant chemotherapy

Exclusion Criteria:

1. Age greater than or equal to 70 years old
2. Abnormal liver and kidney function (more than five times the normal value)
3. Diagnosis level of breast cancer stage 4 or second time tumor patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of tissue distribution of [18F]-DEVD-2 | 7 days
  Biodistribution of [18F] -DEVD-2 evaluated by the maximum standardized uptake value（SUVmax) in various organs during repeated [18F]-DEVD scans will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Chunjing Yu, Principal Investigator — Affiliated Hospital of Jiangnan University
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China